CLINICAL TRIAL: NCT00274300
Title: A Phase I, Two-Center, Open-Label, Dose-Escalating Study to Investigate the Safety, Tolerability and Immunogenicity of pPJV7630, a Therapeutic DNA Vaccine for Herpes Simplex Virus Type 2 (HSV-2), in Patients With Recurrent Genital Herpes Caused by HSV-2
Brief Title: Safety Study of HSV2 DNA Vaccine to Treat Patients With Recurrent Genital Herpes Caused by HSV-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ HSV-001
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2006-01

CONDITIONS: HSV-2
Keywords: DNA vaccine; immunotherapy; Herpes Simplex Virus Type 2 (HSV2); Particle Mediated Epidermal Delivery

INTERVENTIONS:
Biological: pPJV7630 administered by PMED

SUMMARY:
The purpose of this study is to evaluate how well the vaccine is tolerated at sites where administrations are given and any effects it may have on subjects' wellbeing. The study will also test the ability of vaccine to cause particular immune responses in the body and evaluate the effect it has on herpes outbreaks

DETAILED DESCRIPTION:
Herpes simplex virus type 2 (HSV-2) infection is a serious public health problem, with up to 20% of the US population infected. Following primary infection, HSV-2 establishes a latent infection that can lead to recurrent disease when the virus reactivates. Genital lesions are often experienced with viral recurrence and these can be uncomfortable and painful, resulting in significant anxiety and social distress. There are no commercial vaccines available for therapy of HSV-2 infection.The aim of a therapeutic vaccine would be to enhance such natural responses by boosting the appropriate cellular immune response to HSV-2 in those latently infected individuals who experience frequent and unwanted reactivations. The purpose of this study is to evaluate the safety and tolerability profile of the pPJV7630 HSV-2 DNA vaccine as administered by Particle Mediated Epidermal Delivery (PMED )

ELIGIBILITY:
Otherwise healthy subjects with recurrent genital herpes due to HSV-2 infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Adverse Events at all visits
vaccine site evaluations
laboratory parameters pre and post vaccination

SECONDARY OUTCOMES:
HSV recurrences post vaccination
immunogenicity of vaccine post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Larry Stanberry, MD, PhD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Westover Heights Clinic, Portland, Oregon
  - Center for Clinical Studies, Houston, Texas